CLINICAL TRIAL: NCT06311266
Title: Intraoperative Application of a Robot for Endoscopic Neurosurgical Interventions: A Prospective Study
Brief Title: Robotic Endoscopic Neurosurgical Interventions
Acronym: RENI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 34-424 ex 21/22
Record Dates: First submitted 2023-03-29; First posted 2024-03-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Robot for Endoscopic Neurosurgical Interventions
Keywords: robotic; neurosurgery; endoscopic

STUDY DESIGN:
Intervention Model Description: prospective, randomized, single center cohort trial
Who Masked: Participant
Masking Description: Due to the surgical workflow (using the robotic guided device or not) the performing surgical team will not be blinded to the allocated group. However, investigators will be blinded to the allocation of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic (Active Comparator): In the robotic group the endoscope will be guided with the EndoGuide robotic system
  Interventions: Device: Robotic endoscopic neurosurgical intervention
- standard freehand (Active Comparator): In the standard freehand group the endoscope will be guided freehand throughout the surgery
  Interventions: Device: Robotic endoscopic neurosurgical intervention

INTERVENTIONS:
Device: Robotic endoscopic neurosurgical intervention — Robotic guidance device for intraoperative trajectory alignment in endoscopic neurosurgical procedures

SUMMARY:
Endoscopic operations have become increasingly important in the field of neurosurgery over the past decade and require a high degree of precision. Current methods for setting the planned trajectory only offer limited precision due to the manual control, which can lead to complications.

The EndoGuide robot is a modular positioning device for controlling endoscopic instruments, which can use radiological data from neuronavigation to align the trajectory in real time with an accuracy of <0.1mm.

The previous model of the robot is currently approved for interventional radiology and positioning of electrodes and catheters in the field of neurosurgery and is now to be tested in endoscopic neurosurgery.

The investigators therefore expect not only an increase in the accuracy of endoscopic interventions, but also a reduction in morbidity.

DETAILED DESCRIPTION:
Endoscopic procedures, as part of a transnasal pituitary adenoma resection (intervention through the nose to the base of the skull to remove tumors) or ventriculostomy (punctiform opening of a brain chamber to create a bypass circuit for the cerebrospinal fluid), are among the most frequent neurosurgical interventions performed worldwide. The endoscope (ancient Greek: "observe inside") is used for the precise examination of cavities in the context of these minimally invasive interventions. It consists of a rigid tube (diameter approx. 4mm) which transmits the image information of the object or room to be examined through a lens system inside the endoscope shaft to the eyepiece. The light required for the procedure is transmitted from the light source to the tip of the endoscope via the connected light guide, also inside the shaft, through fiber optic bundles.

During neurosurgical interventions, the endoscope is usually guided manually by a second operator. The problem with this manual guidance is the constantly necessary implementation of minimal corrective movements or clouding of the lens due to tissue contact. In case of long lasting interventions, there are also signs of fatigue which lead to unwanted movements of the endoscope. Due to the resulting limited precision and trauma to surrounding tissues, complications and inconclusive results can occur.

In the last 10 years, different surgical devices have been developed to increase procedural accuracy in the field of neurosurgery. For instance, a group presented an automated approach with redundant navigation for minimal invasive extended transsphenoidal skull base surgery successfully performed on cadaveric heads. Furthermore, an assistance system for extended endoscope transsphenoidal skull base surgery has been developed which allowed the simultaneous use of two instruments under endoscopic view. Another approach was to use a force controlled robotic system on bone specimen to increase accuracy for bone milling.

In cooperation with two industrial partners, the COMET Center ACMIT (Austrian Center for Medical Innovation and Technology) developed the MicroMate guidance device that also forms the base for the Stealth AutoGuide system from Medtronic plc. MicroMate is a modular guidance system for surgical invasive tools which provides a precise, submillimetric (<0.1 mm) trajectory alignment according to the predefined navigation data. The setup is based on the iSYS1 robot system, also developed by ACMIT, and on input gained in the course of a clinical trial that has been conducted at the Department of Neurosurgery, Medical University of Vienna 4-10. Notably, none of the two setups mentioned above does impinge on the surgical procedure by itself, nor does it advance any object into the patient. The neurosurgeon remains in control of the instruments during the whole procedure.

The robot used in this study (EndoGuide v2 by ACMIT Gmbh) uses exactly the same mechanical and electronic components as the MicroMate/Stealth AutoGuide system. The only difference between the two CE/FDA certified robots and the EndoGuide platform is a firmware extension to provide a tool pivoting function that allows the endoscope to be rotated around any point along the endoscope shaft. The rotation of the endoscope thus gives the user different views of the area to be viewed.

Aim of the Project The aim of the present study is to evaluate the feasibility and clinical value of the EndoGuide robotic guidance device for intraoperative trajectory alignment in endoscopic neurosurgical procedures (transnasal transphenoidal surgery; ventriculostomy) as compared to the standard freehand method.

With the intraoperative application of the robot the investigators expect:

* an increase in the accuracy of endoscopic interventions and thus a reduction in intervention- related morbidity,
* a reduction in trauma and thus also in secondary bleeding in the context of endoscopic interventions.

Rationale Null hypothesis: There is no significant difference between the accuracy of the endoscopic guidance using the robotic guidance device and the accuracy of the manual method. Primary hypothesis: The intraoperative application of the robotic guidance device for precise trajectory alignment significantly increases the accuracy of navigation-guided endoscopic procedure as compared to the standard manual method and thereby reduces procedure-related morbidity.

1. Hypothesis: The intraoperative application of the robotic guidance device for endoscopic neurosurgical procedures is feasible.
2. Hypothesis: The intraoperative application of the robotic guidance device increases procedural safety.

Objectives Main Objective: Assessment of Target Error as a Measure for Accuracy The target error (TE) measured in mm, corresponds to the distance between the true (surgically performed) trajectory that has been aligned by the robot and the preoperatively defined trajectory stored on the navigation system.

Using fusion of routine pre- and postoperative radiological images, this distance can be calculated with the navigation system software. Study data will be saved in a password-protected data-base only accessible for study personnel.

Secondary Objectives

Additionally to accuracy, the investigators will test for the following measures:

* Rate of procedure-related adverse effects (e.g. hemorrhages)
* Total procedure time (time from skin incision to suture) and setup time (time from positioning the patient to skin incision)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the present study
* Procedure-related patient insurance
* Age 18-80 years
* Diagnosis indicating a ventriculostomy
* Diagnosis of an endo- or suprasellar lesion with indication for transsphenoidal surgery
* MRI and CT scanner compatible

Exclusion Criteria:

* Pregnancy, breast feeding
* Patients not able to reason
* Age <18 or >80 years
* Claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Target Error (TE) | 30 minutes (during procedure)
  Distance in millimeters between the true (surgically performed) trajectory aligned by the robot, and the preoperatively defined trajectory stored on the navigation system.

SECONDARY OUTCOMES:
Adverse Effect | 7 days (through in-patient stay)
  Rate of procedure-related adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bumm K, Wurm J, Rachinger J, Dannenmann T, Bohr C, Fahlbusch R, Iro H, Nimsky C. An automated robotic approach with redundant navigation for minimal invasive extended transsphenoidal skull base surgery. Minim Invasive Neurosurg. 2005 Jun;48(3):159-64. doi: 10.1055/s-2005-870903. PMID 16015493
- [Background] Nimsky Ch, Rachinger J, Iro H, Fahlbusch R. Adaptation of a hexapod-based robotic system for extended endoscope-assisted transsphenoidal skull base surgery. Minim Invasive Neurosurg. 2004 Feb;47(1):41-6. doi: 10.1055/s-2003-812465. PMID 15100931
- [Background] Federspil PA, Geisthoff UW, Henrich D, Plinkert PK. Development of the first force-controlled robot for otoneurosurgery. Laryngoscope. 2003 Mar;113(3):465-71. doi: 10.1097/00005537-200303000-00014. PMID 12616198
- [Background] Fichtinger G, Fiene JP, Kennedy CW, Kronreif G, Iordachita I, Song DY, Burdette EC, Kazanzides P. Robotic assistance for ultrasound-guided prostate brachytherapy. Med Image Anal. 2008 Oct;12(5):535-45. doi: 10.1016/j.media.2008.06.002. Epub 2008 Jun 18. PMID 18650122
- [Background] Korb W, Kornfeld M, Birkfellner W, Boesecke R, Figl M, Fuerst M, Kettenbach J, Vogler A, Hassfeld S, Kornreif G. Risk analysis and safety assessment in surgical robotics: a case study on a biopsy robot. Minim Invasive Ther Allied Technol. 2005;14(1):23-31. doi: 10.1080/13645700510010827. PMID 16754150
- [Background] Schulze F, Buhler K, Neubauer A, Kanitsar A, Holton L, Wolfsberger S. Intra-operative virtual endoscopy for image guided endonasal transsphenoidal pituitary surgery. Int J Comput Assist Radiol Surg. 2010 Mar;5(2):143-54. doi: 10.1007/s11548-009-0397-8. Epub 2009 Sep 4. PMID 20033497
- [Background] Fitzpatrick JM. The role of registration in accurate surgical guidance. Proc Inst Mech Eng H. 2010;224(5):607-22. doi: 10.1243/09544119JEIM589. PMID 20718266
- [Background] Martinez-Moreno M, Widhalm G, Mert A, Kiesel B, Bukaty A, Furtner J, Reinprecht A, Knosp E, Wolfsberger S. A novel protocol of continuous navigation guidance for endoscopic third ventriculostomy. Neurosurgery. 2014 Dec;10 Suppl 4:514-23; discussion 523-4. doi: 10.1227/NEU.0000000000000518. PMID 25121792